CLINICAL TRIAL: NCT03242733
Title: Ultrasound Assessment of Gastric Contents in Fasted Elderly Patients With Hip
Brief Title: Ultrasound Assessment of Gastric Contents in Fasted Elderly Patients With Hip Fracture
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, Associate professor, Department of Anesthesiology and Pain medicine, SMG-SNU Boramae Medical Center
Other Study IDs: 20170804/10/2017/8
Record Dates: First submitted 2017-08-04; First posted 2017-08-08 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Hip Fractures
Keywords: Gastroparesis
MeSH Terms: conditions — Hip Fractures; Gastroparesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hip fracture patients: Fasted elderly patients scheduled for hip fracture surgery except exclusion criteria are enrolled.
  Interventions: Other: Ultrasound assessment of gastric contents

INTERVENTIONS:
Other: Ultrasound assessment of gastric contents — Ultrasound assessment of gastric contents is performed in fasted elderly patients for hip fracture surgery.

SUMMARY:
Evaluation of gastric contents in fasted elderly patients with hip fracture. The gastric contents will be examined by using ultrasonography in fasted elderly patients scheduled for hip fracture surgery. The primary outcome is the number of patients with stomach contents, and the secondary outcome is the component of residual gastric contents.

DETAILED DESCRIPTION:
In the patients who has femur fracture, they are immobilized because of the pain. This condition makes the gastric movement slow, and the pain also contributes to delayed digestion.

In the present study, the gastric content is assessed by using ultrasonography in fasted elderly patients for hip fracture surgery. Ultrasound assessment is performed in the supine position. All patients scheduled elective surgery for hip fracture over 65 years old are objects. The primary outcome is the number of patients with not empty stomach and full stomach, and the secondary outcome is the component of residual gastric contents.

ELIGIBILITY:
Inclusion Criteria:

* Who has hip fracture and agrees with the purpose of the study

Exclusion Criteria:

* gastrointestinal pathology
* history of any type of gastrectomy
* gastrointestinal anomaly

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Who has hip fracture and agrees with the purpose of the study
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-12-26 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Ultrasound assessment of the presence of gastric contents. | Before the induction of anesthesia (Baseline)
  The presence of of gastric contents is assessed by using ultrasonography; yes/no

SECONDARY OUTCOMES:
Ultrasound assessment of the component of residual gastric contents | Before the induction of anesthesia (Baseline)
  The component of residual gastric contents is assessed by using ultrasonography; empty, clear fluid, solid content

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Young Hwang, MD,phD, Study Chair — Seoul National University Boramae Hospital
Locations (1):
- Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Warner MA, Warner ME, Weber JG. Clinical significance of pulmonary aspiration during the perioperative period. Anesthesiology. 1993 Jan;78(1):56-62. doi: 10.1097/00000542-199301000-00010. PMID 8424572
- [Background] Lienhart A, Auroy Y, Pequignot F, Benhamou D, Warszawski J, Bovet M, Jougla E. Survey of anesthesia-related mortality in France. Anesthesiology. 2006 Dec;105(6):1087-97. doi: 10.1097/00000542-200612000-00008. PMID 17122571
- [Background] Landreau B, Odin I, Nathan N. [Pulmonary aspiration: epidemiology and risk factors]. Ann Fr Anesth Reanim. 2009 Mar;28(3):206-10. doi: 10.1016/j.annfar.2009.01.020. Epub 2009 Mar 21. French. PMID 19304443